CLINICAL TRIAL: NCT03335111
Title: The Influence of Bilateral Arm Ischemic Postconditioning on Clinical Prognosis and Outcome in Patients With Acute Ischemic Stroke（BAIPC）
Brief Title: Influence of Bilateral Arm Ischemic Postconditioning on Clinical Prognosis and Outcome in Acute Ischemic Stroke Patients
Acronym: BAIPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BAIPC
Record Dates: First submitted 2017-07-31; First posted 2017-11-07 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Remote Ischemic Postconditioning
Keywords: Remote Ischemic Postconditioning; Peripheral Immunity

STUDY DESIGN:
Intervention Model Description: BAIPC group patients are admistrated by 5 cycles extremities ischemia (5-minute blood-pressure cuff inflation up to 50 mmHg higher than baseline, followed by 5-minute cuff deflation).
Who Masked: Participant
Masking Description: Patients without BAIPC are admistrated by 5 cycles extremities ischemia (5-minute blood-pressure cuff inflation using pressure 0 mmHg , followed by 5-minute cuff deflation). All subjects will take BAIPC for 1 week using 'Remote Ischemic Conditioning Equipment' .
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACI with BAIPC (Experimental): Beside of routine treatment for Anterior circulation infarction(ACI) patients, BAIPC group patients are admistrated by 5 cycles extremities ischemia (5-minute blood-pressure cuff inflation up to 50 mmHg higher than baseline, followed by 5-minute cuff deflation). All subjects will take BAIPC for 1 week using 'Remote Ischemic Conditioning Equipment' .Intravenous blood collection with anticoagulant and 5ml total blood will be administered at 0d, 1d and 7-10d respectively. The blood samples will be stored for laboratory assay. The blood samples only use in this trial.
  Interventions: Procedure: Intravenous blood collection
- ACI without BAIPC (Sham Comparator): ACI patients in this group only recieve routine treatment for ischemic stroke and are admistrated by 5 cycles extremities ischemia (5-minute blood-pressure cuff inflation using pressure 0 mmHg , followed by 5-minute cuff deflation). All subjects will take BAIPC for 1 week using 'Remote Ischemic Conditioning Equipment' .Intravenous blood collection with anticoagulant and 5ml total blood will be administered at 0d, 1d and 7-10d respectively. The blood samples will be stored for laboratory assay. The blood samples only use in this trial.
  Interventions: Other: Remote Ischemic Conditioning Equipment; Procedure: Intravenous blood collection

INTERVENTIONS:
Other: Remote Ischemic Conditioning Equipment — BAIPC is admistrated by 5 cycles extremities ischemia (5-minute blood-pressure cuff inflation up to 50 mmHg higher than baseline, followed by 5-minute cuff deflation) for one week.
  Arms: ACI without BAIPC
Procedure: Intravenous blood collection — Nurses will collect 5 ml intravenous blood with anticoagulant and 5ml total blood at 0d, 1d and 7-10d respectively. The blood samples will be stored for laboratory assay. The blood samples only use in this trial.

SUMMARY:
Influence of bilateral arm ischemic postconditioning （BAIPC）on the injury and protective blood markers and the clinical prognosis and outcome in patients with acute ischemic stroke

DETAILED DESCRIPTION:
In this study, we explore the influence of bilateral arm ischemic postconditioning (BAIPC) to patients with anterior circulation acute ischemic stroke. Patients with anterior circulation acute ischemic stroke are enrolled and divided into control group and experimental group. Patients in experimental group are administrated with BAIPC within 3 days from the occurrence of stroke. The National Institute of Health stroke scale (NIHSS) will be evaluated at different time point to analyze the influence of BAIPC to acute ischemic patients. The level of IL-4, IL-6，TNF-α as well as the frequency of different sub-populations T cells in the blood at different time point will be detected to explore the possible mechanism of BAIPC protective function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ischemic cerebral stroke within 72 hours, NIHSS score between 4 to 15 points;
2. Age between 18-80 years ,gender not limited;
3. freely given informed consent.

Exclusion Criteria:

1. Patients with progressive neurological disease or patients that cannot survive more than 1 year
2. Patients suspected intracranial artery dissection, moyamoya disease, any known vascular inflammatory disease, radioactive vascular lesions, fibromuscular dysplasia, sickle cell disease, tumor, reversible cerebral vascular contraction and reversible posterior leukoencephalopathy syndrome
3. Patients with Cardioembolism , such as rheumatic mitral or aortic stenosis, artificial heart valve, sick sinus syndrome, left atrial myxoma, left ventricular mural thrombus or valvular vegetations, congestive heart failure, bacterial endocarditis
4. Patients with uncontrollable severe hypertension (after drug treatment, systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg) Patients with subclavian artery stenosis 50% or higher or subclavian artery steal blood syndrome and upper limb arterial occlusion
5. Patients with serum Aspertate aminotransferase or Alanine transaminase concentration 3 times higher than normal ceiling Patients that Creatinine clearance < 0.6 ml/s or serum creatinine >265 umol/l (> 3.0 mg/dl)
6. Patients once with intracranial tumors or brain aneurysm, arteriovenous malformation
7. Patients with intracranial bleeding occurred within 90 days (parenchymal hemorrhage, subarachnoid hemorrhage, subdural out/epidural blood), retinal hemorrhage or visceral bleeding occurred within 30 days.
8. Patients with severe blood system disease or severe blood coagulation disfunction , platelet < 100 x 109 / L;
9. Patients that received major surgery 30 days before or is expected to wthin 12 months (including femoral artery, heart, the aorta or the carotid surgery);
10. Patients whose Target lesion blood vessel had received a stent implantation, angioplasty or other medical treatment, or is expected to above treatments witnin 12 months ;
11. Patients with BAIPC contraindications, e.g. severe soft tissue injuries, such as the upper extremity fractures or blood vessels lesions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Changes of pheripheral serum cytokines | 0d, 1d and 7-10d
  We evaluate the changes of the concentration of serum cytokine (IL-4, IL-6, TNF, et.al) at 0d, 1d, 7-10d respectively to demonstrate whether acute stroke would depress the immune state of patients and wether BAIPC can influence the immune state of patients suffering acute stroke.
Changes of pheripheral immune cells | 0d, 1d and 7-10d
  We evaluate the frequency of pheripheral immune cells (Th1, Th2, Th17 and Treg cells) at 0d, 1d and 7-10d to demonstrate whether acute stroke would depress the immune state of patients and wether BAIPC can influence the immune state of patients suffering acute stroke.

SECONDARY OUTCOMES:
Changes of National Institute of Health Stroke scale (NIHSS) | Before BAIPC and after BAIPC for one week
  We evaluate patients NIHSS before BAIPC and after BAIPC for one week to see wether BAIPC could improve the short term prognosis of patient.Scoring Definitions include level of consciousness, visual field, facial palsy,limb motor,sensory ,language,and dysarthria .The NIHSS captures both motor and non-motor impairments of stroke, and provides a good overview of people's deficits.NIHSS ranges from 0 to 42, with high scores corresponding to increased severity of stroke with worse prognosis.
Relapse of ischemic stroke | one year after patients' first stroke
  We observe the relapse of ischemic stroke after one yearto see wether BAIPC could improve the long term prognosis of patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jiachun Feng, MD,Phd, Study Director — The First Hospital of Jilin University
Locations (1):
- First hospital of Jilin University, Changchun, Jilin, China